CLINICAL TRIAL: NCT01202513
Title: Efficacy and Safety of Topical Bimatoprost Solution 0.03% in Stable Vitiligo:A Preliminary Study
Brief Title: Topical Bimatoprost Solution 0.03%in Stable Vitiligo
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: regulatory reasons
Sponsor: Gian Sagar Medical College and Hospital (Other)
Responsible Party: Rajeev Jain, Gian Sagar Medical College and Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GSMCH230810
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2010-07

CONDITIONS: Vitiligo; Repigmentation
Keywords: Vitiligo; Repigmentation
MeSH Terms: conditions — Vitiligo | interventions — Bimatoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bimatoprost application (Experimental)
  Interventions: Drug: Bimatoprost 0.03% topical ophthalmic solution

INTERVENTIONS:
Drug: Bimatoprost 0.03% topical ophthalmic solution

SUMMARY:
Vitiligo is an acquired depigmentation disorder of great cosmetic importance, affecting 1-4% of the world's population. Phototherapy and topical agents such as corticosteroids, calcineurin inhibitors, and vitamin-D derivatives are basic treatment modalities have been used in vitiligo but there is still no effective and safe treatment for this disease. Resistance to therapy, treatment complications and recurrence after treatment are the major problems of the current treatments.

There are no clinical studies of use of Bimatoprost in treatment of vitiligo, as it is supposed to cause more hyperpigmentation and hypertrichosis as compared to other topical prostaglandin analogues; hence, the investigators decided to use it in treatment of localized vitiligo.

DETAILED DESCRIPTION:
Vitiligo is an acquired depigmentation disorder of great cosmetic importance, affecting 1-4% of the world's population. Vitiligo does not cause physical symptoms but because of its unsightly appearance, particularly on dark or tanned skin it can have considerable impact both psychologically and socially. Many ways of restoring normal colour to the skin have been tried but improvement is usually short-lived. The causes of vitiligo are not yet clearly understood, so many treatments have been developed on the basis of limited scientific evidence. There is no cure, and no way of limiting the spread of the disease has so far been found.

The pathogenetic basis of the disease is melanocyte disappearance from achromic patches and experimental evidence has shown that three possible mechanisms enable this to occur: an apoptotic process, a necrotic event, and melanocythoragy following trauma due to impaired function of cell-cell or cell-matrix adhesion.

Prostaglandins (PGs) are biologically active derivatives of 20 carbon atom polyunsaturated essential fatty acids released from cell membrane phospholipids. PGE2 and PGF2 are primary PGs. PGE2 is synthesized in skin and affects keratinocytes, Langerhans cells and melanocytes and regulates melanocyte proliferation. Epidermal melanocytes synthesize melanin in response to ultraviolet radiation (UVR). The mechanisms mediating the UVR-induced activation of melanogenesis are unknown but, as UVR induces the turnover of membrane phospholipids generating prostaglandins (PGs) and other products, it is possible that one of these might provide the activating signal. 1 In an in vitro study by Tomita et al .,2 normal human epidermal melanocytes became swollen and more dendritic when they were cultured with prostaglandin E 2 (PGE 2), but not with PGE 1. In another study by Nordlund et al ., 3 PGE2 applied topically to mice skin caused an increase in melanocyte density.

Histologic studies indicate that PGE 2 also enhances melanogenesis. Recently, there have been many reports of iris darkening, hyperpigmentation of the eyelashes, and periocular hyperpigmentation induced by latanoprost . (prostaglandin F 2 α , used for the treatment of glaucoma). 4,5 Although the exact mechanism of this pigmentation is not clear, different mechanisms of the induction of hyperpigmentation by prostaglandins have been suggested, including: (i) influencing the responsiveness of melanocytes to neuronal stimuli; (ii) causing melanocyte proliferation; and (iii) a direct or second messenger mediated interaction with melanocytes via the stimulation of tyrosinase activity.

Phototherapy and topical agents such as corticosteroids, calcineurin inhibitors, and vitamin-D derivatives are basic treatment modalities have been used in vitiligo but there is still no effective and safe treatment for this disease. Resistance to therapy, treatment complications and recurrence after treatment are the major problems of the current treatments.

There are no clinical studies of use of Bimatoprost 0.03% in treatment of vitiligo, as it is supposed to cause more hyperpigmentation and hypertrichosis as compared to other topical prostaglandin analogues, hence, we decided to use it in treatment of localized vitiligo.

Aim:

In this study, twenty patients with vitiligo will be treated with topical Bimatoprost o.o3% ophthalmic solution for 4 months to elucidate its efficacy and tolerability in stable vitiligo.

Patients and methods In this prospective, interventional, non-randomised, single blind, controlled study, twenty patients with stable vitiligo will be enrolled from the Dermatology out patient department of Gian Sagar Medical College and Hospital. The protocol will follow the Declaration of Helsinki and prior approval of Institutional Review Board will be obtained. Informed consent will be obtained from all patients. Detailed history and physical examination will be obtained. The age, sex, previous treatments, family history, type of vitiligo, durations of disease (in month), areas of involvement, Koebner phenomenon, leukotrichia will be recorded in special data sheet. The diagnosis of vitiligo will be made clinically. No concomitant treatment will be allowed and a washout period of at least 1 month will be given in patients using other therapies.

Patients will be instructed to apply a Bimatoprost 0.03% solution twice daily to the depigmented skin taking care of no spillage to surrounding skin. The dimensions of the treated lesions will be measured in transverse and longitudinal axes at the time of enrollment, subsequently every month till 4 months.

The measurement of the lesions will be performed by an independent observer who is blind to the treatment options. Photography will be done using a digital camera (Sony Digital Still Camera Cyber-shot ModelNO DSCF 717, Tokyo, Japan) at the baseline and at every follow up visit. Patients will be evaluated by the same observer who was blind to the treatment options.

Primary Outcome Measures:

The percentage of repigmentation in the previously depigmented patch, in form of color or size changes and folliculocentric repigmentation, of the treated and the control patches.6

Depending on the extent of repigmentation, the response to the treatment will be graded as:

* no and minimal (<25%),
* moderate (25-49%),
* marked (50-74%),
* excellent (75-99%), and
* complete (100%) response. Response without reduction of the surface and only with perifollicular hyperpigmentation will be categorized as perifollicular pigmentation. Responding lesions will be defined as patches that achieved more than 50% repigmentation as compared with the baseline. Treatment will be discontinued if patients did not show any improvement or worsening at 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of either sex and at least 10 years old
2. Have a diagnosis of vitiligo with no news lesions or growth of old lesions in the past 6 months
3. Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form
4. Agree to follow and undergo all study-related procedures

Exclusion Criteria:

1. Patients showing evidence of spontaneous repigmentation in any of the lesions
2. Patients with rapidly progressive disease were also excluded.
3. Patients with hypersensitivity to the drug or any of its constituents
4. Patients with BSA > 5%

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
repigmentation in the previously depigmented patch | 4 months

SECONDARY OUTCOMES:
safety profile of Topical Bimatoprost solution | 4 month
  Hyperpigmentation of surrounding skin, Allergic reaction to bimatoprost, Hypertrichosis

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Jain, M.D., Study Director — PP; Tarun Narang, MD, Principal Investigator — GSMCH

REFERENCES:
- [Background] Friedmann PS, Wren FE, Matthews JN. Ultraviolet stimulated melanogenesis by human melanocytes is augmented by di-acyl glycerol but not TPA. J Cell Physiol. 1990 Feb;142(2):334-41. doi: 10.1002/jcp.1041420216. PMID 2303529
- [Background] Nordlund JJ, Collins CE, Rheins LA. Prostaglandin E2 and D2 but not MSH stimulate the proliferation of pigment cells in the pinnal epidermis of the DBA/2 mouse. J Invest Dermatol. 1986 Apr;86(4):433-7. doi: 10.1111/1523-1747.ep12285717. PMID 3528310
- [Background] Wand M, Ritch R, Isbey EK Jr, Zimmerman TJ. Latanoprost and periocular skin color changes. Arch Ophthalmol. 2001 Apr;119(4):614-5. No abstract available. PMID 11296032
- [Background] Prota G, Vincensi MR, Napolitano A, Selen G, Stjernschantz J. Latanoprost stimulates eumelanogenesis in iridial melanocytes of cynomolgus monkeys. Pigment Cell Res. 2000 Jun;13(3):147-50. doi: 10.1034/j.1600-0749.2000.130305.x. PMID 10885672
- [Background] Hossain D. Assessment scale used in vitiligo. J Am Acad Dermatol. 2005 Jun;52(6):1110-1. doi: 10.1016/j.jaad.2004.02.028. No abstract available. PMID 15928648
- [Background] Tomita Y, Iwamoto M, Masuda T, Tagami H. Stimulatory effect of prostaglandin E2 on the configuration of normal human melanocytes in vitro. J Invest Dermatol. 1987 Sep;89(3):299-301. doi: 10.1111/1523-1747.ep12471536. PMID 3305717